CLINICAL TRIAL: NCT02675348
Title: Effects of Meat Protein Administration on Body Composition, Strength, Muscle Structure, Immunological and Haematological Markers in Endurance Athletes
Brief Title: Beef Protein Supplementation in Endurance Athletes
Acronym: Beef
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Responsible Party: Principal Investigator, Fernando Naclerio, Principal Lecturer, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fES-uREC-15-1 3 02
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dietary Modification
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dietary Supplement: Beef Protein (Experimental): All the groups will perform a similar endurance training involved 4 to 6 workout per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity. Training session will last from 45 min to a maximum of 120 min.
  Intervention will last for 10 weeks. Participants will ingest 20g of beef protein powder mixed with 250ml of water at post workout (training days) or before breakfast (non training days).
  Interventions: Dietary Supplement: Dietary Supplement: Beef Protein
- Dietary Supplement: Whey Protein (Experimental): All the groups will perform a similar endurance training involved 4 to 6 workout per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity. Training session will last from 45 min to a maximum of 120 min.
  Intervention will last for 10 weeks. Participants will ingest 20g of whey protein powder mixed with 250ml of water at post workout (training days) or before breakfast (non training days).
  Interventions: Dietary Supplement: Dietary Supplement: whey Protein
- Dietary Supplement: CHO (Active Comparator): All the groups will perform a similar endurance training involved 4 to 6 workout per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity. Training session will last from 45 min to a maximum of 120 min.
  Intervention will last for 10 weeks. Participants will ingest 20g of maltodextrin powder mixed with 250ml of water at post workout (training days) or before breakfast (non training days).
  Interventions: Dietary Supplement: Dietary Supplement: CHO

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Beef Protein — Participants will combine a 10-week periodized and controlled endurance programme with the ingestion of beef protein supplement after training. Measurements pre and post intervention will be endurance performance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes
  Other Names: 100% all beef
  Arms: Dietary Supplement: Beef Protein
Dietary Supplement: Dietary Supplement: whey Protein — Participants will combine a 10-week periodized and controlled endurance programme with the ingestion of whey protein supplement after training. Measurements pre and post intervention will be endurance performance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes
  Other Names: Whey protein powder
  Arms: Dietary Supplement: Whey Protein
Dietary Supplement: Dietary Supplement: CHO — Participants will combine a 10-week periodized and controlled endurance programme with the ingestion of maltdextrin after training. Measurements pre and post intervention will be endurance performance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes
  Other Names: maltodextrin
  Arms: Dietary Supplement: CHO

SUMMARY:
The aim of this project is to investigate the potential benefits of combining a new protein beef hydrolysates extract with a regular endurance training programme on (a) body composition (b) performance (c) muscle structure (d) blood markers of health in athletes. As a second objective the investigators will analyse potential differences obtained from the ingestion of the new hydrolysates beef protein extract compared to the ingestion of others commercially available protein sources such as whey and non protein only carbohydrate contrast nutrients.

DETAILED DESCRIPTION:
This investigation involves a 10 weeks randomised, balanced, double blind parallel group between-subjects design aimed to analyse the effects of combining exercise and a post exercise nutrition strategy (hydrolysates beef protein, whey protein or a isocaloric only carbohydrate placebo) on training outcomes, body composition and blood markers after a period of regular training and feeding intervention. Participants will be divided in three-treatment groups 1) Hydrolysed meat-protein (Beef); 2) Whey (Whey) and 3) non-protein iso-energetic placebo (CHO).

Once considered eligible for the study, and after an initial familiarisation period and baseline tests, participants will be randomly assigned to one of the intervention groups: Beef; Whey and CHO. Each group will follow a 10-week periodised endurance training intervention combined with one of the three specific supplementation treatments (Beef, Whey or CHO). Measurements of blood, body composition, muscle structure and endurance performance will be determined before and after the training intervention.

Once informed consent and health history have been obtained, after the baseline Assessment (t1), participants will divided into three similar profile groups, matched by body mass, age, sex and performance (Vo2max). 1) The Beef protein group (Beef n=12) that will take 20g of hydrolysates beef protein powder and 250 ml of water 2) The whey group (n=12) will take 20 g of whey intact isolate powder mixed with 250 ml of water 3) the contrast group (CHO n=12) that will take an iso-energetic non-protein, only carbohydrate (20 f of maltodextrin plus 250 ml of water) contrast.

Participants: Thirty six participants, recruited from Kent, Medway University Campus, will take part in the project. After being informed of all risk, discomforts, and benefits involved, participants will sign a written informed consent regarding their participation.

Intervention Familiarization period: Participants will undertake 1 sessions of familiarisation with the testing procedure. A qualified conditioning coach will control and assists participants in order to guarantee a correct understanding of the assessment procedure (Body composition, vo2max test, muscle thickness, etc). All participants will be instructed about the appropriate use of the Rate of Perceived Exertion (6-20) Borg scale and the heart rate monitor to control the load and training intensity during test and training.

Endurance Training: Participants will commit to follow a polarised triphasic endurance-training model. This model contains three intensity zones calculated as low intensity [≥ the first ventilatory threshold (VT1), ~ 70% HRmax]; moderate intensity [between VT1 and respiratory compensation point or ventilatory threshold 2 (VT2), >70 < 90% HRmax]; and high intensity [>VT2, 90% HRmax] (Esteve-Lanao et al., 2007). Participants will train 4 to 6 times per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity.

Supplementation protocol: Training days: Immediately (<10 min) after com Non-training days: before breakfast.

Supplements and placebo will be provided in powder form and should be mixed with 250 ml of plain water at the moment of consumption. Supplements and placebo will looks and tastes identical.

Thus, a total of one 20g doses will be administered on daily bases. Participants should ingest a total of 70 doses for a total of 10 weeks of study intervention.

Supplement will be provided in 14 days based by a blind researcher after Participants should return back the empty bag of the supplement/placebo consumed during the previous 14 days period.

ELIGIBILITY:
Inclusion Criteria:

* regularly trained endurance athletes,
* aged 30 to 60 years old,
* minimum 2 years of experience,
* volunteers,

Exclusion Criteria:

* any musculoskeletal injuries, metabolic conditions, or diseases;
* use of medications, smoking, and nutritional supplements known to affect physical performance, muscle damage or recovery process (e.g., creatine, whey protein, and amino acids) within 6 weeks prior to the start of the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Body composition | 10 weeks
  Fat-Free mass
Body composition | 10 Weeks
  Fat mass
Muscular thickness | 10 weeks
  vastus medialis thickness
Endurance Performance | 10 weeks
  Vo2max
Endurance Performance | 10 Weeks
  Ventilatory threshold 2
Blood Markers | 10 weeks
  haemoglobin
Blood Markers | 10 weeks
  red blood cell
Blood Markers | 10 weeks
  haematocrit
Blood Markers | 10 weeks
  transferrin

SECONDARY OUTCOMES:
Immunology markers | 10 weeks
  neutrophils
Immunology markers | 10 weeks
  lymphocyte
Immunology markers | 10 weeks
  monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, Ph D, Study Director — University of Greenwich
Locations (1):
- Department of Life and Sports Science, Chatham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes